CLINICAL TRIAL: NCT06098690
Title: Implementing Innovative and Strategic Approaches to Prevent and Mitigate the Deleterious Effects of HPV Across the Lifespan of Hispanics of Mexican Origin: Community Intervention
Brief Title: Culturally Tailored HPV Psychoeducational Multimedia Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas, El Paso (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Eva Moya, Principle Investigator, University of Texas, El Paso
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 8321-2; 2U54MD007592-26 (NIH)
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2024-12

CONDITIONS: Health Knowledge, Attitudes, Practice; Vaccine-Preventable Diseases; Intention; Adherence, Patient
Keywords: Human Papillomavirus Vaccination; Human Papillomavirus Cancer Screening; HPV Cancer Prevention; HPV Cancer Mitigation; Sexual and Reproductive Health; U.S.-Mexico Border Health; Behavioral Research; Community Engaged Research; Health Disparities; Health Inequities; Social Determinants of Health; Male; Female; Adult; Young Adult
MeSH Terms: conditions — Behavior; Vaccine-Preventable Diseases; Patient Compliance; Coitus

STUDY DESIGN:
Intervention Model Description: A parallel trial design will be used to examine the effectiveness of the Culturally Tailored HPV Psychoeducational Multimedia Community Intervention. Community members who are HPV vaccine naïve or under-vaccinated (given vaccine recommendations) will be randomly assigned to one of two conditions: 1) experimental condition in which they receive the tailored multimedia intervention, and 2) active control condition in which they receive general/standard materials.
Who Masked: Participant, Outcomes Assessor
Masking Description: * Participants [blinding]: participants will be randomly assigned to treatment and control groups, they will not be made aware of other participant's receipt of treatment or control materials. Participants will be asked not to discuss this project outside of the intervention; delivery of the intervention or other educational materials will be virtual, limiting the ability of participants to interact with one another during the study.
  * Outcome assessor [blinding]: to reduce bias in the implementation and assessment of the clinical trial, participant information and pre-post survey responses will be maintained separately from the assignment and delivery of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): A tailored HPV psychoeducational multimedia intervention
  Interventions: Behavioral: Culturally Tailored Multimedia Psychoeducational HPV Intervention
- Active Control (Active Comparator): General/standard multimedia materials on HPV and HPV vaccine
  Interventions: Behavioral: General HPV Multimedia Psychoeducational Control Group

INTERVENTIONS:
Behavioral: Culturally Tailored Multimedia Psychoeducational HPV Intervention — The culturally tailored multimedia psychoeducational intervention will involve audio and visual content and will be delivered in a bilingual fashion (English and Spanish) among adults 18-45 years-old.
  Arms: Treatment
Behavioral: General HPV Multimedia Psychoeducational Control Group — The general/publicly available multimedia intervention will involve audio and visual content and will be delivered in a bilingual fashion (English and Spanish) among adults 18-45 years-old.
  Arms: Active Control

SUMMARY:
Community members ages 18 - 45 years old from the El Paso, Texas, U.S.-Mexico Border Region will be recruited to compare psychoeducational multimedia interventions focused on the human papillomavirus (HPV). Our hypothesis is that adults who view culturally tailored multimedia stories encouraging HPV vaccination will report higher vaccine uptake rates.

DETAILED DESCRIPTION:
A sample of vaccine-naive (unvaccinated or under-vaccinated) adult community members ages 18 - 45 years old from the El Paso, Texas, U.S.-Mexico Border Region, will be recruited to participate in a human papillomavirus (HPV) multi-media intervention. Hypothesis: Vaccine-eligible adults who view culturally tailored multimedia stories encouraging HPV vaccination will report significantly stronger vaccine intentions and, subsequently, significantly higher vaccine uptake rates when compared to vaccine-eligible adults exposed to a standard HPV vaccination fact sheet and generic HPV vaccine videos.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages 18 and 45 years old
* Adults who have not completed the HPV vaccine series (unvaccinated or under-vaccinated)
* Adults currently living or working in El Paso County, Texas

Exclusion Criteria:

* Adults who participated in Phases I or II of the larger research project [cross-sectional phases]
* Adults younger than 18 years of age
* Adults older than 45 years of age
* Adults that do not reside, plan to live or work in El Paso County, Texas, within the next 12 months after the start of the intervention
* Adults who are unable to participate in the full study intervention and follow-up time-points
* Adults who cannot complete study participation and activities in either the English or Spanish languages.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Between-group changes in proportions from baseline scores on the Vaccination Decision Stage scale and post-intervention scores of the Community Intervention Survey. | Baseline (pre-assessment), immediately post-intervention (0 months), 1 month post-intervention
  3-item Vaccination Decision Stage scale (HPV vaccine uptake [yes, no], HPV vaccine intention [scored on a likert scale from 1) Strongly disagree to (5) Strongly agree]).

SECONDARY OUTCOMES:
Between-group changes in proportions from baseline scores on the HPV Vaccine Attitudes scale and post-intervention scores of the Community Intervention Survey. | Baseline (pre-assessment), immediately post-intervention (0 months), 1 month post-intervention
  11-item HPV Vaccine Attitudes scale (perceived safety, perceived harm, perceived effectiveness) scored on a Likert scale from Strongly disagree (1) to Strongly agree (5).
Between-group changes in proportions from baseline scores on the HPV Knowledge scale and post-intervention scores of the Community Intervention Survey. | Baseline (pre-assessment), immediately post-intervention (0 months), 1 month post-intervention
  14-item HPV Knowledge scale scored as True (1) or False (0) on a composite average and multiplied by 100 to obtain a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Moya, PhD, LMSW, Principal Investigator — The University of Texas at El Paso, Border Biomedical Research Center
Locations (1):
- The University of Texas at El Paso, Border Biomedical Center, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Collected deidentified individual participant data (IPD), all IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Approximately, starting 6 months-post scholarly publication of previously listed primary and secondary study outcome(s).
Access Criteria: Collected deidentified IPD and supporting information will be provided on a case by case basis following a formal request to the University of Texas at El Paso (UTEP) Institutional Review Board (IRB) and subsequent approval by the Principal Investigator.
URL: http://www.utep.edu/orsp/human-subjects-research/index.html

REFERENCES:
- See also: NIH RePORTER for 2U54MD007592-26 8321 — http://reporter.nih.gov/project-details/9828289